CLINICAL TRIAL: NCT00081419
Title: Timing of Voluntary Movement in Patients With Tourette Syndrome and Chronic Tic Disorder Using EEG and Surface EMG
Brief Title: Timing of Voluntary Movement in Patients With Tourette Syndrome and Chronic Tic Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040153; 04-N-0153
Record Dates: First submitted 2004-04-10; First posted 2004-04-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-12

CONDITIONS: Tourette Syndrome; Tic Disorders
Keywords: Bereitschaftspotential; Timing of Volition; Urge; Conscious Will; Libet's Clock; Tourette Syndrome; Tic Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

SUMMARY:
This study will examine how the brain controls movement in people with Tourette syndrome and chronic tic disorder to determine if the timing of movement is important in whether someone feels "in control" of their movements. Although movements in tic disorders are often characterized as "involuntary," some patients claim that these movements are made voluntarily, or they are unable to decide if they are voluntary or involuntary. Previous experiments have shown that when people are asked to look at a clock and report the time they first decide to make a movement they report times later than the first brain waves associated with movement appear. When they are asked to report the time they first initiate the movement, they report times before the muscles actually begin to move. This study may help determine how the sense of willing and initiating an action is altered in patients with Tourette syndrome and chronic tic disorder, and how people may feel more or less "in control" of their movements.

Normal volunteers and patients with Tourette syndrome or chronic tic disorder between 18 and 65 years of age may be eligible for this study. Control subjects must not have any neurological or psychological disorders, and patients with Tourette syndrome of chronic tic disorder must not have any other neurological disorders. Patients with attention deficit hyperactivity disorder (ADHD) may not enroll in this study.

All participants will have a medical history, physical examination, and a test to determine their level of attention. Patients will be interviewed about their symptoms and complete psychiatric rating scales. In addition, all participants will undergo the following procedures:

Electric shock

Participants look at a clock on a computer screen, the hands of which revolves quickly. While looking at the clock, each participant will be given small, non-painful electric shocks and asked, according to the clock, to say when they received the shocks. The shocks are repeated 40 times.

Arm movement

Participants are asked to lift their arms off a table repeatedly, at random times, while they look at the computer clock. This exercise is repeated 80 times. Of these 80, participants are asked 10 times consecutively to say the time they first had the desire to move their arm, and then 10 consecutively the time they first felt that they were moving their arm.

Electroencephalography (EEG) and Electromyography (EMG)

Participants undergo EEG and EMG durin...

DETAILED DESCRIPTION:
OBJECTIVES: The purpose of this study is to determine how the subjective sense of willing and initiating an action is altered in patients with Tourette Syndrome and Chronic Tic Disorder. Although many definitions of the disease include the characterization of tics as 'involuntary', some patients claim that these movements are voluntarily made, or are unable to decide if they are voluntary or involuntary. Recent studies have shown that the time order in which someone wills a voluntary movement and begins that movement is central to the subjective sense of causality. We propose to examine tics as well as normal, voluntary movements in patients with Tourette Syndrome and Chronic Tic Disorder to identify the time course between the decision to move and the onset of movement. Using Libet's paradigm, we intend to have subjects watch a fast-rotating clock to report the times associated with willing (time W) and initiating (time M) movement; we will also determine electroencephalographic/electromyographic (EEG/EMG) measures of movement.

STUDY POPULATION: We intend to study adult patients with a Diagnostic and Statistical Manual of Mental Disorders diagnosis of a tic disorder and frequent tics as well as normal, healthy volunteers as controls.

DESIGN: We will ask tic patients to rate the "voluntariness" of their tics using a rating scale. We will ask tics patients to look at a fast-rotating clock on a computer screen and note when their movements were willed (time W) and were initiated (time M), for tics as well as normal voluntary movements. Patients will also report the time of a somatosensory stimulus. Surface EMG will determine the time of actual movement, and EEG will record brain potentials associated with movement. The design will be the same for the normal volunteers with the exception that the volunteers will not complete rating scales and will not be experiencing tics.

OUTCOME MEASURES: The primary outcome measure of this study is the latency of times W and M (before EMG onset) in tics patients as correlated with the voluntariness the patients associate with their tics, compared to the time W and M reported for normal voluntary movements in the normal volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Tic Patients:

Patients will be men or women, ages 18-65, with a DSM-IV-TR diagnosis of TS or CTD. Patients will be screened in the NINDS Movement Disorders Outpatient Clinic, and will have neurological and physical examinations. They will be asked to abstain from alcohol and any medications for 24 hours before the study. All subjects participating in the studies will have a valid Clinical Center Medical Record Number.

Normal Volunteers:

Twenty-six normal controls will be included; controls will be screened in the NINDS Movement Disorders Outpatient Clinic, and will have neurological and physical examinations. They will be asked to abstain from alcohol and any medications for 24 hours before the study. All subjects participating in the studies will have a valid Clinical Center Medical Record Number.

EXCLUSION CRITERIA:

Patients younger than 18 years old or older than 65 years old will be excluded from the study.

Tic Patients:

Patients with neurological disorders other than TS or CTD

Patients with Attention deficit hyperactivity disorder (ADHD)

Patients who are not able to abstain from alcohol or medication affecting the central nervous system for 24 hours before the study

Patients not capable of giving an informed consent

Normal Subjects:

Patients with neurological disorders or ADHD

Patients who are not able to abstain from alcohol or medication affecting the central nervous system for 24 hours before the study

Patients not capable of giving an informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2004-04-08; Study Completion 2009-01-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Berardelli A, Curra A, Fabbrini G, Gilio F, Manfredi M. Pathophysiology of tics and Tourette syndrome. J Neurol. 2003 Jul;250(7):781-7. doi: 10.1007/s00415-003-1102-4. PMID 12883917
- [Background] Goetz CG, Leurgans S, Chmura TA. Home alone: methods to maximize tic expression for objective videotape assessments in Gilles de la Tourette syndrome. Mov Disord. 2001 Jul;16(4):693-7. doi: 10.1002/mds.1159. PMID 11481693
- [Background] Gomes G. Problems in the timing of conscious experience. Conscious Cogn. 2002 Jun;11(2):191-97. doi: 10.1006/ccog.2002.0550. PMID 12191936